CLINICAL TRIAL: NCT00948129
Title: Project ACTION: Adult Smoking Cessation Treatment Through Innovative Outreach to Neighborhoods
Brief Title: Mobile Smoking Cessation Intervention in Enhancing Cancer Outreach in Low-Income Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-0336; NCI-2018-00260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0336 (Other: M D Anderson Cancer Center); R01CA141628 (NIH)
Record Dates: First submitted 2009-07-14; First posted 2009-07-29 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cigarette Smoker; Current Every Day Smoker
MeSH Terms: interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (standard care) (Active Comparator): Participants undergo standard of care smoking cessation intervention consisting of brief advice to quit smoking, NRT, and self-help written materials.
  Interventions: Other: Laboratory Biomarker Analysis; Behavioral: Smoking Cessation Intervention
- Group II (enhanced care) (Experimental): Participants undergo standard of care smoking cessation intervention as in Group I and attend a health feedback counseling session at baseline. Participants also receive access to a smoking cessation hotline telephone number and supportive text messages daily for 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Behavioral: Smoking Cessation Intervention; Other: Tobacco Cessation Counseling
- Group III (intensive care) (Experimental): Participants undergo standard of care smoking cessation intervention as in Group I and attend a health feedback counseling session at baseline. Participants also receive access to a smoking cessation hotline telephone number, supportive text messages daily for 12 weeks, and a smoking cessation telephone call over 15 minutes weekly for 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Behavioral: Smoking Cessation Intervention; Behavioral: Telephone-Based Intervention; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Behavioral: Smoking Cessation Intervention — Undergo standard of care smoking cessation intervention
  Other Names: Smoking and Tobacco Use Cessation Interventions
Behavioral: Telephone-Based Intervention — Undergo telephone based smoking cessation intervention
  Arms: Group III (intensive care)
Other: Tobacco Cessation Counseling — Undergo smoking cessation counseling
  Arms: Group II (enhanced care); Group III (intensive care)

SUMMARY:
This trial studies how well a mobile smoking cessation intervention works in enhancing cancer outreach in low-income adult smokers. Mobile smoking cessation intervention may help smokers quit or cut back on smoking, and help increase the range of cancer prevention services provided to low-income adult smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the efficacy of three smoking cessation interventions targeting community based low-income uninsured and underinsured individuals in a group-randomized trial.

II. Evaluate the role of quit motivation, nicotine withdrawal, risk perception, self-efficacy, social support, and negative affect as potential mediators of smoking abstinence.

III. Compare the cost-effectiveness of the three treatment conditions.

OUTLINE: Participants are randomized to 1 of 3 groups.

GROUP I (STANDARD CARE): Participants undergo standard of care smoking cessation intervention consisting of brief advice to quit smoking, nicotine replacement therapy (NRT), and self-help written materials.

GROUP II (ENHANCED CARE): Participants undergo standard of care smoking cessation intervention as in Group I and attend a health feedback counseling session at baseline. Participants also receive access to a smoking cessation hotline telephone number and supportive text messages daily for 12 weeks.

GROUP III (INTENSIVE CARE): Participants undergo standard of care smoking cessation intervention as in Group I and attend a health feedback counseling session at baseline. Participants also receive access to a smoking cessation hotline telephone number, supportive text messages daily for 12 weeks, and a smoking cessation telephone call over 15 minutes weekly for 12 weeks.

After completion of study, participants are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least 100 cigarettes in lifetime
* English or Spanish speaking
* Currently smoking at least 5 cigarettes a day, on average
* Willing to set a quit smoking date within a week of the enrollment

Exclusion Criteria:

* Positive history of a medical condition that precludes use of the nicotine patch
* Current use of nicotine replacement therapy (NRT)
* Current use of other smoking cessation medications (e.g., Chantix or Zyban)
* Pregnant or nursing
* Enrolled in another smoking cessation study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2009-08-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence rate | At 12 months
  The primary method of analysis will be mixed-model logistic regression.
Cost-effectiveness | At 12 months
  Will perform an incremental cost-effectiveness analysis by comparing the expected economic costs and clinical benefits of the three strategies. Will create a decision-analytic model using TreeAge Pro 2007 software to conduct the incremental cost-effectiveness analysis.

SECONDARY OUTCOMES:
Salivary cotinine levels | At 12 months
  Salivary cotinine will be measured using the NicAlert test system.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Vidrine DJ, Frank-Pearce SG, Vidrine JI, Tahay PD, Marani SK, Chen S, Yuan Y, Cantor SB, Prokhorov AV. Efficacy of Mobile Phone-Delivered Smoking Cessation Interventions for Socioeconomically Disadvantaged Individuals: A Randomized Clinical Trial. JAMA Intern Med. 2019 Feb 1;179(2):167-174. doi: 10.1001/jamainternmed.2018.5713. PMID 30556832
- [Derived] Daly AT, Deshmukh AA, Vidrine DJ, Prokhorov AV, Frank SG, Tahay PD, Houchen ME, Cantor SB. Cost-effectiveness analysis of smoking cessation interventions using cell phones in a low-income population. Tob Control. 2019 Jan;28(1):88-94. doi: 10.1136/tobaccocontrol-2017-054229. Epub 2018 Jun 9. PMID 29886411
- [Derived] Vidrine DJ, Fletcher FE, Danysh HE, Marani S, Vidrine JI, Cantor SB, Prokhorov AV. A randomized controlled trial to assess the efficacy of an interactive mobile messaging intervention for underserved smokers: Project ACTION. BMC Public Health. 2012 Aug 25;12:696. doi: 10.1186/1471-2458-12-696. PMID 22920991

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT00948129/Prot_SAP_000.pdf